CLINICAL TRIAL: NCT06706609
Title: Classification of Adult-onset Diabetes in Five Subgroups in Pakistani Population
Status: Not yet recruiting | Type: Observational
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: GTZ-DM-008-24
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus Type 1 and 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to classify adult-onset diabetes patients into distinct data-driven clusters, such as severe insulin-deficient, severe insulin-resistant, mild obesity-related, and mild age-related diabetes, based on clinical and biochemical characteristics. Using a cross-sectional design, data will be collected from individuals attending outpatient diabetes clinics at tertiary care hospitals in Pakistan. The study will analyze the distribution of metabolic and demographic characteristics within each cluster and assess subgroup-specific risks for diabetic complications. Additionally, the relationship between clustering variables and the risk of complications will be evaluated to enhance the understanding of diabetes heterogeneity and its impact on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders whose age of disease onset was older than 16 years
* Patients newly diagnosed with or previously diagnosed with T2D
* Able and willing to provide written informed consent and to comply with the study

Exclusion Criteria:

* Patients with other medical comorbidities (not a complication of diabetes), such as malignancies.
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of adult patients diagnosed with diabetes who are receiving care at endocrinology clinics across Pakistan. Participants will be recruited from outpatient diabetes clinics during their routine visits. The population represents a diverse group of individuals from various socioeconomic and demographic backgrounds, reflecting the heterogeneity of diabetes presentation in the region
Sampling Method: Non-Probability Sample
Enrollment: 394 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Classify patients into data-driven clusters (e.g., severe insulin-deficient, severe insulin-resistant, mild obesity-related and mild age-related diabetes). | At the time of clinic visit during enrollment

SECONDARY OUTCOMES:
Analyze the distribution of metabolic and demographic characteristics within each cluster. | At the time of clinic visit during enrollment
• Assess subgroup-specific risks for diabetic macrovascular complications such as CVD, Stroke/TIA, and microvascular complications such as nephropathy, retinopathy, peripheral and autonomic neuropathy | At the time of clinic visit during enrollment
Evaluate the relationship between clustering variables and complications. | At the time of clinic visit during enrollment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy JC, Matthews DR, Hermans MP. Correct homeostasis model assessment (HOMA) evaluation uses the computer program. Diabetes Care. 1998 Dec;21(12):2191-2. doi: 10.2337/diacare.21.12.2191. No abstract available. PMID 9839117
- [Background] Slieker RC, Donnelly LA, Fitipaldi H, Bouland GA, Giordano GN, Akerlund M, Gerl MJ, Ahlqvist E, Ali A, Dragan I, Festa A, Hansen MK, Mansour Aly D, Kim M, Kuznetsov D, Mehl F, Klose C, Simons K, Pavo I, Pullen TJ, Suvitaival T, Wretlind A, Rossing P, Lyssenko V, Legido-Quigley C, Groop L, Thorens B, Franks PW, Ibberson M, Rutter GA, Beulens JWJ, 't Hart LM, Pearson ER. Replication and cross-validation of type 2 diabetes subtypes based on clinical variables: an IMI-RHAPSODY study. Diabetologia. 2021 Sep;64(9):1982-1989. doi: 10.1007/s00125-021-05490-8. Epub 2021 Jun 10. PMID 34110439
- [Background] Li PF, Chen WL. Are the Different Diabetes Subgroups Correlated With All-Cause, Cancer-Related, and Cardiovascular-Related Mortality? J Clin Endocrinol Metab. 2020 Dec 1;105(12):dgaa628. doi: 10.1210/clinem/dgaa628. PMID 32893854
- [Background] Bonora E, Trombetta M, Dauriz M, Travia D, Cacciatori V, Brangani C, Negri C, Perrone F, Pichiri I, Stoico V, Zoppini G, Rinaldi E, Da Prato G, Boselli ML, Santi L, Moschetta F, Zardini M, Bonadonna RC. Chronic complications in patients with newly diagnosed type 2 diabetes: prevalence and related metabolic and clinical features: the Verona Newly Diagnosed Type 2 Diabetes Study (VNDS) 9. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001549. doi: 10.1136/bmjdrc-2020-001549. PMID 32819978
- [Background] Ahlqvist E, Storm P, Karajamaki A, Martinell M, Dorkhan M, Carlsson A, Vikman P, Prasad RB, Aly DM, Almgren P, Wessman Y, Shaat N, Spegel P, Mulder H, Lindholm E, Melander O, Hansson O, Malmqvist U, Lernmark A, Lahti K, Forsen T, Tuomi T, Rosengren AH, Groop L. Novel subgroups of adult-onset diabetes and their association with outcomes: a data-driven cluster analysis of six variables. Lancet Diabetes Endocrinol. 2018 May;6(5):361-369. doi: 10.1016/S2213-8587(18)30051-2. Epub 2018 Mar 5. PMID 29503172
- [Background] Anjana RM, Baskar V, Nair ATN, Jebarani S, Siddiqui MK, Pradeepa R, Unnikrishnan R, Palmer C, Pearson E, Mohan V. Novel subgroups of type 2 diabetes and their association with microvascular outcomes in an Asian Indian population: a data-driven cluster analysis: the INSPIRED study. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001506. doi: 10.1136/bmjdrc-2020-001506. PMID 32816869
- See also: Sample Size Calculator — https://www.openepi.com/SampleSize/SSPropor.htm
- See also: Magliano DJ, Boyko EJ; IDF Diabetes Atlas 10th edition scientific committee. IDF DIABETES ATLAS [Internet]. 10th edition. Brussels: International Diabetes Federation; 2021. Chapter 3, Global picture. — https://www.ncbi.nlm.nih.gov/books/NBK581940/